CLINICAL TRIAL: NCT01033682
Title: Evaluation of Bladder Volumes in Patients Receiving Radiotherapy to the Rectum, Using Kilovoltage Cone-beam Imaging
Acronym: FILL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Dr Diana A. Tait, Royal Marsden NHS Foundation Trust
Other Study IDs: CCR3175
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to implement and access a newly developed bladder filling protocol for patients receiving radiotherapy for rectal cancer using imaging on the treatment unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving radical radiotherapy to rectal malignancies.
* Age > 18 years old
* No previous lower GI radiotherapy
* Written informed consent according to good clinical practice (GCP) and national / local regulations.

Exclusion Criteria:

* Patients receiving palliative radiotherapy to rectal malignancies.
* Patients receiving radical short course preoperative radiotherapy for rectal malignancies.
* Patients unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving radiotherapy to the rectum
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who are able to achieve a bladder volume within +/- 30% of planning volume, on all treatment CBCT (cone beam computed tomography) scans

SECONDARY OUTCOMES:
The per-patient standard deviation of bladder volume throughout the course of radiotherapy
The percentage of patients who are unable to follow the bladder filling protocol at any point during their treatment.
The correlation between bladder volume and small bowel volume planning target volume

CONTACTS AND LOCATIONS:
Overall Officials: Dr Diana Tait, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom